CLINICAL TRIAL: NCT04478175
Title: Prospective Evaluation of a Program for Early Identification of Needs and Multidisciplinary Intervention in Supportive Care in Digestive Oncology - DISSPO Parcours Dig' Study
Brief Title: Prospective Evaluation of a Program for Early Identification of Needs and Multidisciplinary Intervention in Supportive Care in Digestive Oncology
Acronym: DParcoursDig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2020-01
Record Dates: First submitted 2020-07-01; First posted 2020-07-20 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Non-colorectal Cancer (Esophagus, Stomach, Liver/Bile Ducts, Pancreas, Neuroendocrine Carcinoma); Colorectal With Associated Risk Factors
Keywords: advanced gastrointestinal (GI) cancers
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced gastrointestinal (GI) cancers (Other): All patients will receive usual care including:
  * Chemotherapy at the investigator's choice,
  * Outpatient clinical visits according to the regular schedule,
  * Tumor evaluation based on tumor marker serum levels, as appropriate, and TAP-CT with intravenous contrast injection every 8 weeks.
  Nutritional support will consist of:
  * A nutrition assessment by a dieticianat W4 and W8 (plus additional visits if required),
  * Nutritional intervention ± oral supplementation, enteral tube feeding, and/or parenteral nutrition).
  Physical activity support will consist of:
  * A physical condition assessment by a APA profesional including physical tests (6-minute walking test, handgrip test, chair stand fitness test, get-up and go test, balance in single-leg and bipodal stance) at baseline, W4 and W8,
  * Personalized counselling for unsupervised home-based exercises
  Interventions: Other: multidisciplinary assessment and intervention

INTERVENTIONS:
Other: multidisciplinary assessment and intervention — early multidisciplinary assessment and intervention in addition to usual patient care

SUMMARY:
Patients with advanced gastrointestinal (GI) cancers are very often sarcopenic/malnourished at diagnosis (> 60% of cases) and at high risk of rapid clinical deterioration. These patients have important supportive care needs that represent a major challenge for improving treatment tolerance and patient survival and health-related quality of life (HRQoL).

Malnutrition and sarcopenia (muscle wasting and dysfunction) are associated with an increased risk of death, complications from chemotherapy, infections, emergency procedures and hospitalizations, and increased costs of care. Therefore, malnutrition and sarcopenia represent a major clinical target in GI cancers.

Interventions targeting malnutrition/sarcopenia should be implemented as early as possible in patients' pathways, these syndromes being reversible at early stages but not at late stages.

A multidisciplinary assessment at diagnosis and therapeutic approach combining nutritional support and and adapted physical activity (APA) in addition to anticancer treatments should be systematically implemented in patients with advanced GI cancers.

This type of intervention complies with the standards recommended by the National Cancer Institute (INCa) to promote the practice of physical activity during and after treatment in oncology.

DETAILED DESCRIPTION:
All patients will receive usual care including:

* Chemotherapy at the investigator's choice,
* Outpatient clinical visits according to the regular schedule,
* Tumor evaluation based on tumor marker serum levels, as appropriate, and TAP-CT with intravenous contrast injection every 8 weeks.

Nutritional support will consist of:

* A nutrition assessment by a dietician including a VAS of food intakes at baseline, at W4 and W8 (plus additional visits if required),
* Nutritional intervention according to the Société Francophone de Nutrition Clinique et Métabolisme (SFNEP) guidelines (dietetic counseling for all patients ± oral supplementation, enteral tube feeding, and/or parenteral nutrition).

Physical activity support will consist of physical condition assessed by International Physical Activity Questionnaire (IPAQ), performance status (ECOG PS), resting heart rate and blood pressure, 6-minute walking test (speed, fatigue), handgrip test, chair stand fitness test, get-up and go test, balance in single-leg and bipodal stance.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Age ≥ 18 years (no superior limit),
3. Histologically confirmed (1) non-colorectal cancer (esophagus, stomach, liver/bile ducts, pancreas, neuroendocrine carcinoma) or (2) colorectal with associated risk factors i.e. ECOG PS 2 (defining significant limitation in daily activities), and/or weight loss ≥ 5% in 1 month or ≥ 10% in 6 months (defining malnutrition/HAS 2019),
4. Advanced disease not amenable to surgery, radiation, or combined modality therapy with curative intent (previous resection of primary tumor allowed), treated with first-line chemotherapy for advanced disease (previous [neo]adjuvant chemo[radio]therapy allowed); or resectable/potentially resectable disease receiving a triplet chemotherapy regimen in a peri-operative setting (e.g. FOLFIRINOX, FLOT) (moderate risk at frailty score)
5. Patients able to attend for administration of chemotherapy,
6. Life expectancy ≥ 3 months,
7. Registration in a National Health Care System (Couverture Maladie Universelle [CMU] included).

Exclusion Criteria:

1. Other active non gastro-intestinal cancers
2. Any medical (including psychiatric, musculoskeletal, or neurological) condition contra-indicating exercise practice,
3. Pregnancy or breastfeeding,
4. Protected adults (individuals under guardianship by court order).

Note: participation to another concomitant clinical trial is allowed, but the patient must inform the Investigator and get an authorization from the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Program faisability | 12 months
  Program feasibility will be satisfactory if ≥ 80% of patients with advanced GI cancers included in the program complete the baseline, W4 and W8 assessments

SECONDARY OUTCOMES:
Dimensions of EORTC QLQ-C30 | 12 months
  EORTC QLQ-C30 completion
Fatigue measured by Visual Analogue Scale (VAS) | 12 months
  Visual Analogue Scale (VAS) completion, a score form 0 to 10 will be given
Pain measured by VAS and analgesics consumption | 12 months
  VAS completion and analgesics consumption report, a score form 0 to 10 will be given and report of analgesics consumption will be given by name and dose
Nutritional status/inflammation measure | 12 months
  weight in kilograms, body mass index will be reported in BMI in kg/m^2, food intakes
Physical condition assessed | 12 months
  International Physical Activity Questionnaire (IPAQ),
Geriatric assessment if age ≥ 70 | 12 months
  G8 score from 0 to 17
Chemotherapy tolerance assessed | 12 months
  toxicities (using Common Terminology Criteria for Adverse Events [CTCAE v5.0])
Progression Free Survival and Overall Survival | 12 months
  Progression Free Survival and Overall Survival
Patient's satisfaction measured by VAS | 12 months
  VAS completion with a score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Véronique GILLON, Study Chair — Institut Curie
Locations (1):
- Institut Curie, Paris, France